CLINICAL TRIAL: NCT04154943
Title: A Phase 2 Study of Neoadjuvant Cemiplimab for Stage II to IV (M0) Cutaneous Squamous Cell Carcinoma (CSCC)
Brief Title: Study of Cemiplimab in Patients With Type of Skin Cancer Stage II to IV Cutaneous Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1901; 2019-003007-35 (EudraCT Number); 2022-500811-37-00 (EU CTIS Number)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: CSCC; Stage II; Stage III; Stage IV; CSCC of Head/neck; CSCC of Extremity; CSCC of Trunk
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab (Experimental): Will receive IV infusion Q3W
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: REGN2810; Libtayo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of neoadjuvant cemiplimab as measured by Pathologic complete response (pCR) rate per independent central pathology review.

The secondary objectives of the study are:

* To evaluate the efficacy of neoadjuvant cemiplimab on measures of disease response, including:
* Major pathologic response (mPR) rate per independent central pathology review
* pCR rate and mPR rate per local pathology review
* ORR prior to surgery, according to local assessment using RECIST 1.1
* To evaluate the efficacy of neoadjuvant cemiplimab on event free survival (EFS), disease free survival (DFS), and overall survival (OS)
* To evaluate the safety profile of neoadjuvant cemiplimab
* To assess change in surgical plan (ablative and reconstructive procedures) from the screening period to definitive surgery, both according to investigator review and independent surgical expert review
* To assess change in post-surgical management plan (radiation, chemoradiation, or observation) from the screening period to post-surgery pathology review, both according to investigator review and independent surgical expert review

ELIGIBILITY:
Key Inclusion Criteria

* Stage II to IV (M0) CSCC, for which surgery would be recommended in routine clinical practice. For stage II patients, lesion must be ≥3 cm at the longest diameter.
* At least 1 lesion that is measurable by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ, bone marrow function, and hepatic function as defined in the protocol

Key Exclusion Criteria

* Solid malignancy within 5 years of the projected enrollment date, or hematologic malignancy (including chronic lymphocytic leukemia [CLL]) at any time
* Distant metastatic disease (M1), visceral and/or distant nodal
* Prior radiation therapy for CSCC
* Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of the first dose of study drug.
* Patients with active, known, or suspected autoimmune disease that has required systemic therapy within 5 years of the projected enrollment date.
* History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HBV or HCV) infection; or diagnosis of immunodeficiency
* Active tuberculosis

NOTE: Other protocol-defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (21):
- United States (14):
  - Regeneron Study Site, Palo Alto, California
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Omaha, Nebraska
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Durham, North Carolina
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
- Australia (3):
  - Regeneron Study Site, St Leonards, New South Wales
  - Regeneron Study Site, Herston, Queensland
  - Regeneron Study Site, Melbourne, Victoria
- Germany (4):
  - Regeneron Study Site, Dresden
  - Regeneron Study Site, Essen
  - Regeneron Study Site, Kiel
  - Regeneron Study Site, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Gross ND, Miller DM, Khushalani NI, Divi V, Ruiz ES, Lipson EJ, Meier F, Su YB, Swiecicki PL, Atlas J, Geiger JL, Hauschild A, Choe JH, Hughes BGM, Schadendorf D, Patel VA, Homsi J, Taube JM, Lim AM, Ferrarotto R, Yoo SY, Mathias M, Han H, Seebach F, Lowy I, Fury MG, Rischin D. Neoadjuvant cemiplimab and surgery for stage II-IV cutaneous squamous-cell carcinoma: follow-up and survival outcomes of a single-arm, multicentre, phase 2 study. Lancet Oncol. 2023 Nov;24(11):1196-1205. doi: 10.1016/S1470-2045(23)00459-X. Epub 2023 Oct 21. PMID 37875144
- [Derived] Gross ND, Miller DM, Khushalani NI, Divi V, Ruiz ES, Lipson EJ, Meier F, Su YB, Swiecicki PL, Atlas J, Geiger JL, Hauschild A, Choe JH, Hughes BGM, Schadendorf D, Patel VA, Homsi J, Taube JM, Lim AM, Ferrarotto R, Kaufman HL, Seebach F, Lowy I, Yoo SY, Mathias M, Fenech K, Han H, Fury MG, Rischin D. Neoadjuvant Cemiplimab for Stage II to IV Cutaneous Squamous-Cell Carcinoma. N Engl J Med. 2022 Oct 27;387(17):1557-1568. doi: 10.1056/NEJMoa2209813. Epub 2022 Sep 12. PMID 36094839

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As of the data cutoff (01 Dec 2021), 101 participants were screened for study eligibility. 79 participants were randomized and received at least 1 dose of cemiplimab.
Groups:
- Cemiplimab 350mg Q3W: Participants received cemiplimab, administered at a dose of 350mg every 3 weeks for up to 4 doses
Period: Overall Study
Arm/Group | Cemiplimab 350mg Q3W
Started | 79
Completed | 0
Not Completed | 79
Not completed — Study Ongoing | 68
Not completed — Lost to Follow-up | 1
Not completed — Decision by the Investigator | 1
Not completed — Death | 5
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  17 years and under | 0
  18 to 64 years | 18
  65 to 84 years | 54
  85 years and over | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 69
    Asian | 1
    Other | 1
    Unknown / Not Reported | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Not Hispanic or Latino | 74
    Unknown/Not Reported | 5

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Major Pathologic Response (mPR) as Assessed by Independent Central Pathology Review
Time Frame: Up to 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants | 10

2. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR) as Assessed by Independent Central Pathology Review
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants | 40

3. Secondary Outcome: Number of Participants With Pathologic Complete Response (pCR) as Assessed by Local Pathology Review
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants | 42

4. Secondary Outcome: Number of Participants With Major Pathologic Response (mPR) as Assessed by Local Pathology Review
Time Frame: Up to 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants | 10

5. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) Prior to Surgery, According to Investigator Assessment Using RECIST 1.1
Time Frame: Up to 12 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Percentage of Participants | 68.4 [56.9 to 78.4]

6. Secondary Outcome: Number of Participants With Planned and Actual Surgery After Neoadjuvant Cemiplimab
Time Frame: Up to 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants
  Participants with Planned Mohs Surgery | 2
  Participants with Actual Mohs Surgery | 2
  Participants with Planned Non-Mohs Surgery | 77
  Participants with Actual Non-Mohs Surgery | 68

7. Secondary Outcome: Number of Participants With Planned and Actual Post-Surgical Management
Time Frame: Up to 14 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350mg Q3W
Number analyzed (Participants) | 79
Participants
  Planned radiation therapy after surgery | 47
  Actual radiation therapy after surgery | 17

8. Secondary Outcome: Event Free Survival (EFS)
Time Frame: Up to 50 Months
Reporting Status: Not Posted, anticipated posting 2026-09

9. Secondary Outcome: Disease Free Survival (DFS)
Time Frame: Up to 47 Months
Reporting Status: Not Posted, anticipated posting 2026-09

10. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 50 Months
Reporting Status: Not Posted, anticipated posting 2026-09

11. Secondary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Up to 52 Months
Reporting Status: Not Posted, anticipated posting 2026-09

12. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Time Frame: Up to 52 Months
Reporting Status: Not Posted, anticipated posting 2026-09

13. Secondary Outcome: Incidence of Deaths
Time Frame: Up to 52 Months
Reporting Status: Not Posted, anticipated posting 2026-09

14. Secondary Outcome: Incidence of Laboratory Abnormalities
Time Frame: Up to 52 Months
Reporting Status: Not Posted, anticipated posting 2026-09

ADVERSE EVENTS:
Time Frame: From first dose to the end of treatment period (Week 25) up to 01-DEC-2021 Data cut-off
Groups:
- Cemiplimab 350 mg Q3W: Participants received cemiplimab, administered at a dose of 350mg every 3 weeks for up to 4 doses
Arm/Group | Cemiplimab 350 mg Q3W
All-Cause Mortality (participants affected / at risk) | 6/79
Serious Adverse Events (participants affected / at risk) | 15/79
Other Adverse Events (participants affected / at risk) | 60/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W (N=79)
Myocardial infarction (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W (N=79)
Diarrhoea (Gastrointestinal disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 10 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5)
Fatigue (General disorders) | 24 (29)
Pyrexia (General disorders) | 4 (5)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT04154943/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04154943/SAP_001.pdf